CLINICAL TRIAL: NCT00590681
Title: Avastin and Temozolomide Following Radiation and Chemotherapy for Newly Diagnosed Glioblastoma Multiforme: A Phase II Study
Brief Title: Bevacizumab and Temozolomide Following Radiation and Chemotherapy for Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15149A
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one (Experimental): This is an open-label, single arm, multi-center, phase II study involving 48 subjects with newly diagnosed supra-tentorial GBM. Following surgery, subjects with radiographically evaluable disease will receive external beam radiotherapy (59.4 - 60 Gy in 30 - 33 fractions) with daily temozolomide (75 mg/m2). Two to three weeks later, subjects will begin treatment with temozolomide (150-200 mg/m2 daily for five of 28 consecutive days) in conjunction with Avastin (10 mg/kg, every 14 days).
  Interventions: Drug: Bevacizumab and Temozolomide

INTERVENTIONS:
Drug: Bevacizumab and Temozolomide — This is an open-label, single arm, multi-center, phase II study involving 48 subjects with newly diagnosed supra-tentorial GBM. Following surgery, subjects with radiographically evaluable disease will receive external beam radiotherapy (59.4 - 60 Gy in 30 - 33 fractions) with daily temozolomide (75 mg/m2). Two to three weeks later, subjects will begin treatment with temozolomide (150-200 mg/m2 daily for five of 28 consecutive days) in conjunction with Avastin (10 mg/kg, every 14 days).
  Other Names: Avastin

SUMMARY:
This study is being conducted to help determine whether the addition of Avastin (an anti-cancer drug), when given along with temozolomide during the monthly cycles that follow radiation, is able to delay tumor growth, shrink tumors, or impact how long people with GBM live. This study is sponsored by Genentech, Inc., the manufacturer of Avastin.

Avastin is the experimental drug being administered in this research study. Avastin binds a protein called vascular endothelial growth factor, or VEGF. VEGF is produced by tumors and circulates in the blood. One of VEGF's main roles is to support the growth of new blood vessels. During cancer, VEGF promotes the growth of blood vessels that bring nutrients to tumor cells and help them grow. Avastin binds to VEGF, which then prevents VEGF from functioning. In laboratory studies, Avastin prevented the growth of several different types of cancer cells grown in animals. Avastin was approved by the Food and Drug Administration (FDA) for the treatment of metastatic colorectal cancer in combination with chemotherapy. Avastin has not been approved by the FDA for the treatment of GBM and is, therefore, considered experimental. Avastin is currently undergoing testing (alone and in combination with another anti-cancer drug, irinotecan) in persons with GBM that have come back after conventional treatment.

Temozolomide (Temodar) is an anti-cancer drug that works by interfering with the growth of cells (including cancer cells) by stopping their division. Temozolomide was approved by the U.S. FDA for the treatment of newly diagnosed GBM in 2005.

Avastin and temozolomide are currently being used together in several research studies involving people with newly diagnosed GBM. Limited information is available about either the safety or effectiveness of this drug combination.

DETAILED DESCRIPTION:
The study consists of the following: 1) a screening period of up to 28 days; 2) a treatment period of radiation with daily temozolomide that lasts approximately 6 weeks, 3) a study treatment period that will last until either your tumor grows or you experience unacceptable side effects; and 4) a 30-day follow-up period after treatment has ended. Additionally, basic information concerning your condition will be collected every 2 months after the follow-up period for the rest of your life.

During this study, Dr. Nicholas and his research team will collect information about you for the purposes of this research. This includes name, address, dates (i.e., date of birth, date of consent), telephone number, and medical record number. Slides of your tumor tissue that were used to diagnose your GBM will be sent to a pathologist to confirm the diagnosis of GBM. After this review has been completed your slides will be returned to the hospital that provided them. Preserved samples of your tumor will also be sent for a test to determine how effective the temozolomide might be in your case. Any remaining tissue will be returned to the hospital that provided it.

Screening phase (following diagnosis of GBM at surgery) To determine if you are eligible to participate in this study, you will undergo a screening process that will involve the following

* Assessment of your cancer by magnetic resonance imaging (MRI) of your brain using an intravenous (in your vein) contrast material
* Recording of your general medical, surgical and cancer history
* Physical examination, including measurement of your blood pressure, height and weight
* Evaluation of your performance status (your ability to carry on daily activities)
* Neurologic examination (how well your nerves and muscles work)
* Blood sample for laboratory tests (approximately 2 to 3 tablespoons) to evaluate your blood counts, liver, and kidney function
* Serum pregnancy test if you are a woman of childbearing potential
* Urine sample
* Recording of any medications taken within the past 14 days

Radiation and daily temozolomide chemotherapy You will begin radiation treatment within 5 weeks of surgery. You will take temozolomide orally once daily (seven days a week) during radiation treatments (which occur Monday - Friday and last approximately six weeks). You will take a medication to prevent a rare form of pneumonia (pneumocystis carinii) that can occur when temozolomide is given on a daily basis. That may be either in pill form or inhaled. During radiation treatment you will be seen every two weeks by a study doctor at which time you will be asked how you are tolerating the treatment. A physical examination, (including neurological evaluation), will be performed. Blood tests (1-2 tablespoons) will be performed to assure that you are not having any side-effects from the chemotherapy.

Post-radiation treatment Two to four weeks after completing radiation you will have a brain MRI scan. Beginning four weeks after radiation ends, the study drug and temozolomide will begin. The study drug (Avastin) will be administered by IV infusion (through a vein) every 2 weeks. Temozolomide will be taken orally for five consecutive days of every 28 days. In other words, you will receive two intravenous infusions of Avastin and five days of temozolomide every 28 days. This constitutes a treatment cycle. These cycles will continue indefinitely. The dose of Avastin will be based upon your weight during screening and will remain the same throughout the study. The temozolomide dose during radiation will be based on your height and weight at screening. During the study phase, temozolomide will be dosed according to your height and weight at the beginning of each treatment cycle. The dose may be delayed for up to four weeks if your blood counts are low. If temozolomide still cannot be given because your blood counts are low for longer than four weeks, the temozolomide will be stopped but the Avastin may still be continued.

Your first dose of Avastin will be given as over 90 minutes. If you tolerate the 90 minute infusion well, infusions in the future may be given over a shorter period of time. However, if you do not tolerate the shorter infusion time, future infusions will be given over the longer period that you previously tolerated. If you experience any problems during or following the infusion, you will be monitored by trained staff until it is considered safe for you to leave.

The dose of Avastin that you receive may be stopped or slowed based on how well you tolerate the treatment. If you must stop treatment because of unfavorable side effects, you may be able to restart treatment once the side effect has improved or resolved. Your doctor will discuss with you whether it is in your best interest to continue treatment. If you stop study drug treatment, you should continue to return to be evaluated as explained below.

Temozolomide will be taken at bedtime on an empty stomach (at least 2 hours after any meal). Prior to each dose of temozolomide, you will take an anti-nausea pill (ondansetron, granisetron, or dolasetron) to reduce nausea and vomiting.

The treatment cycles described above will continue until: 1) your tumor grows, 2) you have unacceptable side effects, 3) you choose to withdraw from this research study, or 4) your participation is ended by Dr. Nicholas or Genentech.

During the first treatment day of each 28 day cycle you will receive Avastin. Your blood pressure will be monitored, and you will have a physical examination, a neurologic examination, and an evaluation of your performance status (how well you are functioning in daily activities). On the same day, you will begin temozolomide chemotherapy. You will have a blood sample drawn for laboratory tests (approximately 2-3 tablespoons), and a urine sample taken. You will be asked by the study doctor about any health problems you have and medications you take. Additional blood samples may be drawn at the discretion of your doctor as part of your standard care.

On day 14 of every treatment cycle you will return to the clinic to receive an infusion of Avastin. At that time, your blood pressure will be taken, and you will have a physical examination and an evaluation of your performance status. On day 21 of each cycle you will have blood work (1-2 tablespoons) to see how well you are tolerating the treatment. Every 8 weeks (after every 2 cycles immediately prior to your next cycle) you will have an MRI of your brain to determine measurements of your tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Disease-Specific Concerns Histologically confirmed GBM as determined by central pathology review Supratentorial location
2. General Medical Concerns 18 years of age; Karnofsky performance status > 60; Tumor-related contrast enhancement on initial and post-operative Gd-MRI; Recovery from effects of surgery and/or its complications prior to initiating radiotherapy; Radiotherapy must begin < 5 weeks following surgery; Pre-and post-operative Gd-MRI prior to the initiation of radiotherapy; Adequate hematological, renal, and hepatic function:hemoglobin > 10 grams hematocrit > 30%, platelets > 100,000 per mm3, BUN < 25 mg/dl, Creatinine < 1.5 mg/dl, Total bilirubin < 1.5 mg/dl, SGOT or SGPT < twice institutional normal range, Subjects must not be pregnant or nursing, Use of effective means of contraception (men and women) in subjects of child-bearing (women) and at all ages (men), Study-specific signed informed consent, Ability to comply with study follow-up procedures.

   -

Exclusion Criteria:

* a. Disease-Specific Concerns: malignant gliomas graded less than GBM; infratentorial tumor location; recurrent disease; intra-tumoral hemorrhage; Placement of Gliadel® wafers; b. Bevacizumab-Specific Concerns: Inadequately controlled hypertension (defined as systolic blood pressure 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications); Any prior history of hypertensive crisis or hypertensive encephalopathy; History of myocardial infarction or unstable angina within 6 months prior to study enrollment; History of stroke or transient ischemic attack within 6 months prior to study enrollment; New York Heart Association (NYHA) Grade II or greater CHF (see Appendix E); Significant vascular disease (e.g., aortic aneurysm, aortic dissection); Symptomatic peripheral vascular disease; Evidence of bleeding diathesis or coagulopathy; History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment; History of intracerebral abscess within 6 months prior to study enrollment; Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment (exclusive of craniotomy); anticipation of need for major surgical procedure during the course of the study; Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment; Serious non-healing wound, ulcer, or bone fracture; Proteinuria at screening as demonstrated by either; Urine protein:creatinine (UPC) ratio 1.0 at screening OR Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible); Known hypersensitivity to any component of Avastin. c. General Medical Exclusions

Subjects meeting any of the following criteria are ineligible for study entry:

Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin cancer study; History of any other malignancy within 5 years (except non-melanoma skin cancer or carcinoma in situ of the cervix);Pregnant or nursing females; Unstable systemic disease, including active infection, uncontrolled hypertension, or serious cardiac arrhythmias requiring medication;

Screening clinical laboratory values:

Absolute neutrophil count < 1500/ul, Platelet count < 100,000/ul, Total bilirubin > 1.6 mg.dl, AST/ALT > 1.5 x the upper limit of normal ( ULN), Creatinine > 1.2 x ULN, Urine protein/creatinine ratio > 1.0, International normalized ration (INR) > 1.5 and activated partial thromboplastin time (aPTT) > 1.5 x ULN (except for subjects receiving anticoagulation therapy) in the absence of therapeutic intent to anticoagulate the subject. Therapeutic anticoagulation is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kelly Nicholas, MD PhD, Principal Investigator — University of Chicago; Martin Kelly Nicholas, MD, PhD, Principal Investigator — University of Chicago
Locations (5):
- United States (5):
  - The University of Chicago, Chicago, Illinois
  - NorthShore University health system, Evanston, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Medical college of Wisconsin, Milwaukee, Wisconsin
  - Waukesha health care, Waukesha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: This is an open-label, single arm, multi-center, phase II study involving 48 subjects with newly diagnosed supra-tentorial GBM. Following surgery, subjects with radiographically evaluable disease will receive external beam radiotherapy (59.4 - 60 Gy in 30 - 33 fractions) with daily temozolomide (75 mg/m2). Two to three weeks later, subjects will begin treatment with temozolomide (150-200 mg/m2 daily for five of 28 consecutive days) in conjunction with Avastin (10 mg/kg, every 14 days).
  Bevacizumab and Temozolomide: This is an open-label, single arm, multi-center, phase II study involving 48 subjects with newly diagnosed supra-tentorial GBM. Following surgery, subjects with radiographically evaluable disease will receive external beam radiotherapy (59.4 - 60 Gy in 30 - 33 fractions) with daily temozolomide (75 mg/m2). Two to three weeks later, subjects will begin treatment with temozolomide (150-200 mg/m2 daily for five of 28 consecutive days) in conjunction with Avastin (10 mg/kg, every 14 days).
Period: Overall Study
Arm/Group | Treatment
Started | 62
Completed | 42 (The forty-two participants who did proceed to the post-RT phase)
Not Completed | 20
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 8
Not completed — Death | 3
Not completed — Lost to Follow-up | 1
Not completed — disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 62
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.4 [55.5 to 66.6]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are 19 patients without gender information.
  Participants
    number analyzed (Participants) | 43
    Female | 19
    Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 56
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: The best clinical response rates determined and 95% confidence intervals obtained using the exact binomial distribution.
Time Frame: Up to 3 years
Population: The forty-two participants did proceed to the post-RT phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 62
percentage of participants
  Complete Response | 22.5 [12.9 to 35.0]
  Partial Response | 19.4 [10.4 to 31.4]
  Stable Disease | 11.3 [4.7 to 21.9]
  Progression | 6.5 [1.8 to 15.7]

2. Primary Outcome: Progression-free Survival (PFS)
Time Frame: Up to 3 years
Population: The forty-two participants did proceed to the post-RT phase, and 60 patients had valid data.
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Treatment
Number analyzed (Participants) | 60
years | 0.96 [0.80 to 1.68]

3. Secondary Outcome: Safety of Avastin in Combination With Temozolomide in This Study Population
Description: Toxicity rates (limited toxicity to grade 4+)
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 62
Participants
  Apnea | 1
  Bone infection | 1
  Creatine phosphokinase increased | 1
  DIC | 1
  Death | 1
  Depression | 1
  Fatigue | 1
  Febrile neutropenia | 1
  Hypocalcemia | 1
  Ischemia cerebrovascular | 1
  Leukocytes | 1
  Leukopenia | 2
  Metabolic | 1
  Musculoskeletal | 1
  Neutrophils | 2
  Platelets | 2
  Pleural effusion | 1
  Proteinuria | 2
  Seizure | 1
  Soft tissue infection | 1
  Thrombosis | 1
  Lymphopenia | 1

4. Secondary Outcome: Duration of Response
Description: Duration of response time from the first assessment of CR or PR until disease progression or death from any cause, whichever occurs first, event-free survival probability at two years assessed by Kaplan-Meier survivor function
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Treatment
Number analyzed (Participants) | 24
probability | 38.8 [19.3 to 58.0]

5. Secondary Outcome: Overall Survival
Time Frame: Up to 3 years
Population: The forty-two participants did proceed to the post-RT phase, and 60 patients had valid data.
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Treatment
Number analyzed (Participants) | 60
years | 1.68 [1.28 to 2.31]

6. Secondary Outcome: Changes in Relative Cerebral Blood Volume (rCBV) of Tumors After (2 Infusions) of Avastin
Time Frame: Up to 3 years
Population: Zero participants were analyzed due to no data.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 3/62
Other Adverse Events (participants affected / at risk) | 53/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=62)
Anorexia (Metabolism and nutrition disorders) | 1
Seizure (Nervous system disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=62)
Abdominal pain (Gastrointestinal disorders) | 5
Alanine aminotransferase (Investigations) | 15
Alkaline phosphatase (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 34
Anorexia (Metabolism and nutrition disorders) | 17
Aspartate aminotransferase increased (Investigations) | 9
Auditory/Ear (Ear and labyrinth disorders) | 6
Blood bicarbonate decreased (Investigations) | 5
Bruising (Injury, poisoning and procedural complications) | 6
Confusion (Psychiatric disorders) | 9
Constipation (Gastrointestinal disorders) | 27
Constitutional Symptoms (General disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Cushingoid (Endocrine disorders) | 7
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 18
Diarrhea (Gastrointestinal disorders) | 15
Dizziness (Nervous system disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Ear, nose, and throat examination abnormal (Investigations) | 7
Edema (General disorders) | 14
Fatigue (General disorders) | 46
Fever (General disorders) | 5
Headache (Nervous system disorders) | 24
Heartburn (Gastrointestinal disorders) | 4
Hemoglobin (Investigations) | 18
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 9
Hyperbilirubinemia (Hepatobiliary disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 25
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 15
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypotension (Vascular disorders) | 4
Infection (Infections and infestations) | 4
Insomnia (Psychiatric disorders) | 9
Joint pain (Musculoskeletal and connective tissue disorders) | 13
Depression (Psychiatric disorders) | 7
Leukocytes (Blood and lymphatic system disorders) | 12
Lymphopenia (Blood and lymphatic system disorders) | 29
Memory impairment (Nervous system disorders) | 10
Metabolic/Lab (Metabolism and nutrition disorders) | 6
Muscle weakness (Musculoskeletal and connective tissue disorders) | 17
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 7
Nausea (Gastrointestinal disorders) | 31
Neurological disorder NOS (Nervous system disorders) | 6
Neurology - Other (Psychiatric disorders) | 4
Ocular - Other (Eye disorders) | 4
Pain (General disorders) | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Peripheral sensory neuropathy (Nervous system disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Platelets (Investigations) | 22
Proteinuria (Renal and urinary disorders) | 6
Pulmonary - Other (Infections and infestations) | 6
Rash (Skin and subcutaneous tissue disorders) | 17
Seizure (Nervous system disorders) | 8
Speech disorder (Nervous system disorders) | 4
Taste alteration (Nervous system disorders) | 9
Thrombosis (Vascular disorders) | 5
Tremor (Nervous system disorders) | 6
Upper respiratory infection (Infections and infestations) | 5
Urinary frequency (Renal and urinary disorders) | 8
Urinary tract infection (Infections and infestations) | 5
Vision blurred (Eye disorders) | 5
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 13
Neutrophils (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No